CLINICAL TRIAL: NCT07364630
Title: A Multicenter, Prospective, Controlled Modified Multi-Platform Trial Assessing the Efficacy of Human Placental Membrane Products and Standard of Care in the Management of Nonhealing Diabetic Foot Ulcers and Venous Leg Ulcers.
Acronym: BIORESCUE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: BioLab Holdings (Industry)
Collaborators: Serena Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RescueX
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Diabetic Foot Ulcer; Foot Ulcer Chronic; DFU; Ulcer Foot; Venous Leg Ulcer (VLU); Venous Leg Ulcer; Venous Ulcer; Leg Ulcers; Ulcer
Keywords: Leg Ulcer; Ulcer; Venous Ulcer; Venous Leg ulcer; VLU; DFU; Diabetic Foot Ulcer; Foot Ulcer; Diabetic foot
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Varicose Ulcer; Leg Ulcer; Ulcer

STUDY DESIGN:
Intervention Model Description: This study follows a rescue design: patients in the SOC arm who fail to heal during the BIOCAMP Prospective Modified Dual Platform Multicenter Randomized Controlled Clinical Trial will enter the Rescue trial and receive one of the study products.
  Patients enrolled in this trial must still meet medical necessity criteria for cellular, acellular, matrix-like, products (CAMPs) recently published by the Medicare Administrative Contractor's (MAC) in their local coverage determinations (LCD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Tri-Membrane Wrap™ DFU (Other): Tri-Membrane Wrap™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Tri-Membrane Wrap™ DFU
- Membrane Wrap™ DFU (Other): Membrane Wrap™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap™ DFU
- Membrane Wrap-Lite™ DFU (Other): Membrane Wrap-Lite™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap-Lite™ DFU
- Membrane Wrap-Hydro™ DFU (Other): Membrane Wrap-Hydro™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap-Hydro™ DFU
- Tri-Membrane Wrap™ VLU (Other): Tri-Membrane Wrap™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Tri-Membrane Wrap™ VLU
- Membrane Wrap™ VLU (Other): Membrane Wrap™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap™ VLU
- Membrane Wrap-Lite™ VLU (Other): Membrane Wrap-Lite™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap-Lite™ VLU
- Membrane Wrap-Hydro™ VLU (Other): Membrane Wrap-Hydro™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap-Hydro™ VLU

INTERVENTIONS:
Other: Tri-Membrane Wrap™ DFU — Participants will receive weekly applications of Tri-Membrane Wrap™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Tri-Membrane Wrap™ DFU
Other: Membrane Wrap™ DFU — Participants will receive weekly applications of Membrane Wrap™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Membrane Wrap™ DFU
Other: Membrane Wrap-Lite™ DFU — Participants will receive weekly applications of Membrane Wrap-Lite™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Membrane Wrap-Lite™ DFU
Other: Membrane Wrap-Hydro™ DFU — Participants will receive weekly applications of Membrane Wrap-Hydro™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Membrane Wrap-Hydro™ DFU
Other: Tri-Membrane Wrap™ VLU — Participants will receive weekly applications of Tri-Membrane Wrap™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Tri-Membrane Wrap™ VLU
Other: Membrane Wrap™ VLU — Participants will receive weekly applications of Membrane Wrap™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Membrane Wrap™ VLU
Other: Membrane Wrap-Lite™ VLU — Participants will receive weekly applications of Membrane Wrap-Lite™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Membrane Wrap-Lite™ VLU
Other: Membrane Wrap-Hydro™ VLU — Participants will receive weekly applications of Membrane Wrap-Hydro™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Membrane Wrap-Hydro™ VLU

SUMMARY:
The study is a multicenter, prospective, controlled modified multi-platform trial assessing the efficacy of human placental membrane products and standard of care in the management of nonhealing diabetic foot ulcers and venous leg ulcers.

DETAILED DESCRIPTION:
This study follows a rescue design: patients in the SOC arm who fail to heal during the BIOCAMP Prospective Modified Dual Platform Multicenter Randomized Controlled Clinical Trial will enter the Rescue trial and receive one of the study products.

Patients enrolled in this trial must still meet medical necessity criteria for cellular, acellular, matrix-like, products (CAMPs) recently published by the Medicare Administrative Contractor's (MAC) in their local coverage determinations (LCD).

ELIGIBILITY:
Inclusion Criteria:

* The potential subject must be at least 18 years of age or older.
* The potential subject must have a diagnosis of type 1 or 2 Diabetes mellitus.
* If the potential subject has two or more ulcers, the target ulcer must be the same ulcer treated in the BIOCAMP study.
* The potential subject must consent to using the prescribed offloading method for the duration of the study.
* The potential subject must agree to attend the weekly study visits required by the protocol.
* The potential subject must be willing and able to participate in the informed consent process.
* The potential subject must have participated in the BIOCAMP trial in the SOC only arm and NOT achieved complete closure by the 12-week endpoint.

Exclusion Criteria:

* The potential subject is known to have a life expectancy of < 6 months.
* The potential subject's target ulcer is not secondary to diabetes.
* The target ulcer is infected or there is cellulitis in the surrounding skin.
* The target ulcer exposes tendon or bone.
* There is evidence of osteomyelitis complicating the target ulcer.
* There is an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
* The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
* The potential subject is taking hydroxyurea.
* The potential subject has applied topical steroids to the ulcer surface within one month of TV-1.
* The potential subject with a previous partial amputation on the affected foot that results in a deformity that impedes proper offloading of the target ulcer.
* The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of TV-1.
* The potential subject has an acute Charcot foot, or an inactive Charcot foot, which impedes proper offloading of the target ulcer.
* The potential subject is a woman who is pregnant or considering becoming pregnant within the next 6 months.
* The potential subject has end stage renal disease requiring dialysis.
* The potential subject, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
* The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
* The potential subject did not participate in the BIOCAMP trial.
* The potential subject participated in the BIOCAMP trial and was not randomized to the SOC only arm.
* The potential subject participated in the BIOCAMP trial and achieved complete closure.
* The target ulcer was treated with CAMPs, also defined as skin substitute, or hyperbaric oxygen therapy (HBOT) in the month prior to TV-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Wound Closure | 1-12 Weeks
  The percentage of target ulcers achieving complete wound closure in 12 weeks.

SECONDARY OUTCOMES:
Time to Closure | 1-12 weeks
  Time to closure for the target ulcer.
Percentage Area Reduction | 1-12 weeks
  Percentage wound area reduction from TV-1 to TV-13 measured weekly with digital photographic planimetry, using imaging device, and physical examination.
Adverse Events | 1-12 Weeks
  The number of product- or procedure- related adverse events.
Determine improvement in Quality of Life | 1-12 weeks
  To determine the between-arm difference in the quality of life for subjects receiving HPM plus SOC compared to SOC alone using the Forgotten Wound Score (FWS) questionnaire. Forgotten wound scores situations on a scale of "never" to "mostly."
Determine improvement in Quality of Life | 1-12 weeks
  To determine the between-arm difference in the quality of life for subjects receiving HPM plus SOC compared to SOC alone using the Wound Quality of Life (wQOL) questionnaire. Scores on a scare from "Not at all" to "Very much."
Pain in patients who present with VAS greater than 4 | 1-12 Weeks
  To determine the between-arm difference in pain for patients that present with a Visual Analog Sale (VAS) score of greater than 4. The VAS has a scale of 0-10. 0 Meaning no pain and 10 being the worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Foot and Ankle Disorders, Philidelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No